CLINICAL TRIAL: NCT00614276
Title: TENDRILS: A Multimedia Intervention for Women's Sexual Dysfunction After Cancer
Brief Title: Female Sexual Dysfunction Intervention
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0340
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2013-10

CONDITIONS: Sexual Dysfunction
Keywords: Sexual Dysfunction; Cancer-related Sexual Dysfunction; Female Cancer Survivors; Tendrils; Website program; Self-help tool; Sexual counseling; Questionnaires
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Phase I - Focus Groups
  Interventions: Behavioral: Focus Group; Behavioral: TENDRILS; Behavioral: Questionnaires
- Phase II TENDRILS: Phase II - TENDRILS Program only.
  Interventions: Behavioral: TENDRILS; Behavioral: Questionnaires
- Phase II TENDRILS + Counseling: Phase II - TENDRILS + Sexual Counseling Sessions.
  Interventions: Behavioral: TENDRILS; Behavioral: Questionnaires; Behavioral: Sexual Counseling Sessions

INTERVENTIONS:
Behavioral: Focus Group — To evaluate a multimedia intervention program for women with cancer-related sexual dysfunction.
  Groups: Phase I - Focus Groups
Behavioral: TENDRILS — Tendrils: A Sexual Renewal Program for Women Surviving Cancer - a website designed to give women information about sexual problems related to cancer and its treatment, and the website suggests ways to overcome those problems.
Behavioral: Questionnaires — The questionnaires ask about your background (such as age, education, relationships), your cancer diagnosis and treatment, and the quality of your life in terms of your health, your general emotions, and your sexual function. The questionnaires take about 30-45 minutes to complete.
Behavioral: Sexual Counseling Sessions — Attend 3 sexual counseling sessions at M. D. Anderson.
  Groups: Phase II TENDRILS + Counseling

SUMMARY:
The goal of this psychosocial research study is to learn whether a website program called "Tendrils: Sexual Renewal for Women after Cancer " may help female cancer survivors improve their sex lives when used either as a self-help tool or in combination with brief sexual counseling by a health care professional.

Objectives:

Sexual dysfunction is the most common long-term consequence of cancer treatment, affecting half of survivors of breast and gynecological cancer and many women treated for other cancers. Yet, few women get the help they need for sexual problems. Our primary objective is to develop and evaluate a multimedia intervention program for women with cancer-related sexual dysfunction. Tendrils: A Sexual Renewal Program for Women Surviving Cancer will: 1) explain the causes of cancer-related sexual dysfunction; 2) offer self-help strategies to prevent or overcome problems; 3) advise women on seeking appropriate medical help; and 4) possibly serve as the core of a counseling program, along with a therapist manual. Tendrils is aimed at a wide audience, from newly diagnosed to long-term survivors, across cancer sites. Material will be presented with sensitivity to religious and cultural attitudes about sexuality. Animations will illustrate anatomy and physiology. The software will let women use Tendrils in a variety of formats: over the internet, on a CD-Rom, printed out, or as downloaded digital video or audio on a handheld computer or media player. Video vignettes will illustrate problems and strategies. Five female cancer survivors will host the program, sharing their experiences.

DETAILED DESCRIPTION:
The Tendrils website is designed to give women information about sexual problems related to cancer and its treatment, and the website suggests ways to overcome those problems. The website can be viewed on a computer, or parts of it may be printed out or downloaded to portable media players (such as mp3 players). The program includes videos describing women's personal experiences with sexual problems after cancer.

If you appear to be eligible to take part in this study, you will be mailed an informed consent form to review and sign and a 19-item questionnaire about your sexual function that may take 5 to 10 minutes to complete. If the questionnaire results also show you are eligible for the study, and you have completed the informed consent form, you will be given a user name and password to view the Tendrils web site. On the web site you will fill out a set of questionnaires. The questionnaires ask about your background (such as age, education, relationships), your cancer diagnosis and treatment, and the quality of your life in terms of your health, your general emotions, and your sexual function (such as your desire for sex, ability to enjoy sex, and/or any problems with painful sex). In total, the questionnaires will take about 30-35 minutes to complete. If your questionnaires suggest that you are very depressed or upset, a psychologist on the research team will request an in-person interview with you to discuss your feelings. The psychologist will decide whether taking part in the study would be too stressful for you. If this is the case, you will be taken off study. You will also be given a list of referrals for mental health care in the community.

You will be randomly assigned (as in the toss of a coin) to one of 2 groups. There will be an equal chance of being assigned to either group. If you are assigned to Group 1, you will work with the Tendrils program for 12 weeks on your own. If you are assigned to Group 2, in addition to working with the Tendrils program on your own, you will attend 3 sexual counseling sessions at M. D. Anderson.

Once you have submitted your questionnaires, you will view the Tendrils website over the internet at home over the course of 12 weeks. If you do not log onto the Tendrils website within 2 weeks after receiving your user name and password, you will be called on the telephone as a reminder. If you do not log on within 4 weeks, you will be taken off study and your password will expire.

To use the Tendrils website, you will read the information, listen to audio interviews of women discussing their sexual problems after cancer (or view videotaped interviews), and practice "homework" that is designed to help to improve your sexual life. The women in the videos discuss, for example, the types of sexual problems they had (such as losing the desire for sex or experiencing pain during sex), how their sexual problems affected their self-esteem or relationships, and what the women did to solve the sexual problems. The videos do not show real people having sexual activity.

The homework may involve writing or dictating comments in a section called "My Journey" about how cancer affected your sex life or fertility. This is just for your own private use, unless you choose to share your writing with your counselor. Writing the comments may take about 15-20 minutes each time. The homework may also involve trying what is called "relaxing touch" with your partner, learning to tense and relax muscles around your vaginal entrance, or trying to change negative thoughts about sex. You will be able to use the website on your own schedule, but it is estimated that you may spend 30-60 minutes per week on the website, plus another 30 minutes per week of homework time. The homework may be practiced alone or with your sexual partner. Your partner will be given a separate user name and password to view Tendrils during the 12 weeks. Your partner will not be able to view your comments in "My Journey," or your questionnaires, however.

When you use the Tendrils website, the system will record how many times you visit the website, how much time you spend on each visit, and which web pages you view. Any time you leave the Tendrils website, the recording stops. The recording only happens on the Tendrils website.

Participants assigned to Group 2 will attend 3 sexual counseling sessions at M. D. Anderson during the 12-week study. Each counseling session will last about an hour. The counselor will be a trained health care professional who will try to help you get the most out of the Tendrils program.

Once a week during the 12 weeks, participants in both Group 1 and Group 2 will be asked to log onto the Tendrils website and answer 3 questions about the website. This is called a diary entry. The questions ask how much time you spent reading printouts from the website, listening to audio or viewing video portions of the website on a portable media player, or doing homework recommended on the website.

You will be able to access the website after the 12 weeks, as long as the research study is in progress. However, your password will become inactive if you do not complete questionnaires at the end of 12 weeks.

At the end of the 12 weeks, and then 3 months and 6 months later, you will be asked to complete the same questionnaires that you completed at the beginning of the study. You will not need to answer the medical questions or questions about your background. If the sexual relationship ends during the course of the study, you will still be asked to complete these follow-up questionnaires. You will be able to access the website during the 6-month follow-up period.

If you receive a loaner laptop, you will be asked to return it at the end of the 12 weeks. However, you will still be able to access the website using any computer that has an internet connection, for example at the home of a friend or at a public library. You will also have the option of coming to M. D. Anderson to complete follow-up questionnaires online and we will compensate you for parking.

The Tendrils website is hosted on a secure server, which means that the information you give online is protected by a special firewall. Your user name and password will be different than your real name. No identifying information, such as your real name or address, will be entered in the Tendrils website. Only the study chair and 1 or 2 members of the research team will be able to see the list that links your user name and password to your real name. The list of passwords and names will be destroyed at the end of the project.

After returning the last questionnaire at the 6-month follow-up time, your participation in the research study will be finished.

This is an investigational study. If you do not have a computer, researchers will try to loan you a laptop during the study. (If a loaner laptop is not available, it is possible that you may have to be on a waiting list to start the study until someone else finishes using the laptop.) Postage-paid return envelopes for the questionnaires will be provided, if needed. Loaner printers are available.

Up to 240 women will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I: Woman cancer survivor
2. Phase I: Speaks and reads English well enough to evaluate the website and participate in a focus group
3. Phase II: Had breast cancer or a gynecological cancer diagnosed 1 to 5 years previously
4. Phase II: Has a sexual partner in relationship of at least 6 months' duration.
5. Phase II: Has a score on the Female Sexual Function Inventory below the cut-off criterion indicating sexual dysfunction (i.e. less than 26.55 total score).
6. Phase II: Lives in commuting distance of MDACC so that can attend 3 counseling sessions if randomized to professional treatment group.
7. Phase II: Currently no evidence of active cancer.
8. Phase II: Not receiving any cancer treatment other than hormonal therapy.

Exclusion Criteria:

1. Phase I: Under age 18
2. Phase II: Under age 18
3. Phase II: Currently in mental health care for a sexual problem.
4. Phase II: BSI-18 at study entry indicates high distress and a visit with project staff confirms that the participant is too distressed to benefit safely from the intervention.
5. Phase II: Cannot arrange for participant to have privacy when accessing internet at home, even if we offer loaner laptop and subsidized internet service.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women, over 18 years old, with cancer-related sexual dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2007-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Total score on Female Sexual Function Index (FSFI) | Baseline, after the 12-week treatment period, and at 3- and 6-month follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie R Schover, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org